CLINICAL TRIAL: NCT05571020
Title: Effect of Mat Pilates Exercise on Musculoskeletal System, Body Composition and Psychosocial Status In Healthcare Providers: A Randomised Control Trial
Brief Title: Effect of Mat Pilates Exercise on Musculoskeletal System, Body Composition and Psychosocial Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Collaborators: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Sanem ŞENER, associated professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ZonguldakBEU
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Healthcare Providers; Health-Related Behavior; Exercise
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mat Pilates Group (Experimental): Two days a week, approximately one hour a day, for a total of eight weeks, in groups of 5-6 people, they were included in the mat pilates exercise program.
  Before starting the exercise program, the study group participants were informed about the principles of the pilates working system (I am not sure if this statement is correct terminologically), the training program and the 5 key elements of the pilates approach, neutral spine (head-neck-shoulder-waist-abdominal placement), lumbopelvic stabilization, Informative training on scapular stabilization, focusing and breathing was given.
  Interventions: Other: mat pilates
- Control Group (No Intervention): Control group participants did not participate in any exercise program.

INTERVENTIONS:
Other: mat pilates — Both groups adapted for their rides by not participating in a different exercise and meal. In the study, they were not found in any store in the control groups. In the Mat-Pates Group, information about the 5 key elements of the study and pilates team, perspective (-neck-shoulder-waist-abdominal placement), lumbopel stabilization, scapular stabilization, review and information was covered. Then, in the study groups, it was purchased from groups of 5-6 people at most for one hour a day. In order to participate in all these application activities, he continues his life without participating in any evaluation.
  Arms: Mat Pilates Group

SUMMARY:
The aim of this study is to investigate Mat Pilates exercise on the musculoskeletal system, body composition, and psychosocial status, Fatigue, SeverityScale, sleep quality, mood disorder.

Method: Participants were randomly divided into two groups as Mat-PilatesGroup (n=16) and Control Group (n=16). Mat-PilatesGroup participants were given Mat Pilates exercise for about 1 hour per day, twice a week for 8 weeks, accompanied by a physiotherapist. Control Group participants did not participate in any exercise program.

DETAILED DESCRIPTION:
Healthcare workers constitute a professional group that is physically and mentally burdened. Working in bad posture for long periods of time and being exposed to high occupational psychological stress both cause musculoskeletal pain and pose a high psychological risk. Stress-related risk factors such as standing for a long time at the workplace, insufficient rest times, and a working system in the form of shifts are common.

Because time spent at work covers a large part of the day, it is inevitable that the work environment will have a significant impact on physical, social and psychological health. It is known that group exercises performed with colleagues in the company of a therapist at work are more effective in increasing vitality, improving pain and anxiety control, and increasing commitment to participation in exercise compared to exercise performed at home.Jakopsen et al. examined the effect of workplace-based exercises and home-based exercise in a randomized controlled study that included 200 female health workers working in 18 departments in three different hospitals. They observed that the group participants who exercised at work achieved more positive results in terms of muscle strength, musculoskeletal pain, and use of painkillers than the home-based exercise group.

Pilates method; It is an exercise approach based on the theories of motor learning, core stability and body-mind-spirit interaction with the aim of reducing pain and disability, improving and rehabilitating physical abilities, with principles such as breathing, concentration, centering, control, precision and fluency. Mat-Pilates is the most common type of pilates, which has 2 working styles: Mat-Pilates and instrumented Pilates, and it uses gravity for core stabilization.

The aim of this study; The aim of this study is to investigate the effect of eight-week mat pilates exercises performed with a physiotherapist in the workplace on the musculoskeletal system, body composition and psychosocial status of healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 20-60,
* volunteer to participate in the study, healthcare workers,
* lack of habit of exercising regularly in participants,
* Those who can regularly participate in the exercise program to be applied

Exclusion Criteria:

* have a disease that may prevent them from exercising (cardiovascular, pulmonary and orthopedic),
* having vision and/or hearing loss, pregnancy status,
* a history of loss of balance due to loss of consciousness or dizziness,
* balance disorder due to the diagnosis of peripheral vestibular disease,
* having a pacemaker or metal implant in their body

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
weight in kilograms | Change from Baseline weight in kilograms at 2 months
  evaluated with a bioelectrical impedance analyzer (Tanita RD-545)
height in meters | 2 months
  The height of the participants was measured using a fixed stadiometer with 0.5 cm precision.While the person is standing during the measurement; Measurements were taken without shoes, head upright, feet touching the wall with heels together, knees tense, body upright and head in Frankfort plane.
waist circumference measurement | Change from Baseline waist circumference measurement at 2 months
  Individuals were asked to stand with arms outstretched and feet together, and measurements were taken from the narrowest part of the trunk. Since it is difficult to determine the narrowest part of the trunk in obese individuals, the evaluation was made from the midpoint between the ribs and the iliac crest.
hip circumference measurement | Change from Baseline hip circumference measurement at 2 months
  The widest protrusion level of the hip muscles was measured at the level of the symphysis pubis anteriorly and in the posterior region.
waist/hip ratio circumference measurement | hange from Baseline waist/hip ratio circumference measurement at 2 months
  It was calculated by dividing the waist circumference (cm) of the individuals by the hip circumference (cm). Waist/hip Ratio is the most commonly used anthropometric method to determine fat distribution. While waist circumference of 90 cm and above determines the risk increase in men, this measurement is 80 cm and above in women. Waist circumference of 102 cm or more in men and 88 cm or more in women indicates a significant increased risk for coronary heart disease and metabolic complications.
Body Mass Index | Change from Baseline Body Mass Index at 2 months
  weight and height will be combined to report BMI in kg/m^2)
Body Fat Ratio | Change from Baseline Body Fat Ratio at 2 months
  evaluated with a bioelectrical impedance analyzer (Tanita RD-545)
Fat Mass | Change from Baseline Fat Mass at 2 months
  All carbohydrates, fats and proteins that are in excess of the need in the body turn into adipose tissue. A large part of this transformed warehouse is located under the skin, especially in the thigh, hip and chest area.
bilateral arm circumference measurement | Change from Baseline bilateral arm circumference measurement at 2 months
  The midpoint between the acromion and the olecranon was found and marked on the arm. The individual was asked to stand and flex the elbow by contracting the biceps brachii muscle. Circumference measurement was taken from the widest part of the muscle.
leg circumference measurement | Change from Baseline bilateral leg circumference measurement at 2 months
  The measurement was made in a standing position. Measurements were made at the midpoint between the inguinal region and the proximal part of the patella or where the muscle was most swollen. 10-15 cm above the patella corresponds to this point
Flexibility Assessment | Change from Baseline Flexibility Assessment at 2 months
  Trunk Flexion and Hamstring Length, Trunk Hyperextension, Trunk Lateral Flexion
Psychosocial Status Assessment | Change from Baseline Psychosocial Status Assessment at 2 months
  Quality of Life (Short Form) Scale: The scale includes a total of 36 items and 8 subsections to be answered considering the last four weeks. health status is evaluated between 0 and 100 points in total. 0 indicates worst health, 100 indicates best health.
Fatigue Severity | Change from Baseline Fatigue Severity at 2 months
  Fatigue Severity Scale: The Turkish version of the Fatigue Severity Scale (ref) was used to evaluate the fatigue status of individuals. The scale assesses the state of fatigue in the last four weeks, including the day it was filled. Individuals score between 0 and 7 (for each question?) on the scale, which consists of 9 questions in total. High scores indicate increased fatigue
Sleep Quality | Change from Baseline Sleep Quality at 2 months
  Pittsburg Sleep Quality index: The Turkish version of the Pittsburg Sleep Quality Index (ref) was used for the quantitative evaluation of sleep quality. The scale consists of a total of 24 questions, 19 of which are self-report (self-report) questions and 5 of which are answered by the individual's spouse or roommate (these questions are not included in the calculation), and it evaluates the last one-month period. Self-assessment questions are related to sleep quality and do not indicate sleep disturbance and the prevalence of the disorder. The 18 items scored are grouped into seven component scores (subjective sleep quality, sleep delay, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction). The total score of the seven components is equal to the total index score. Each item is scored between 0-3 and the total score varies between 0-21. A total score of five or more indicates poor sleep quality.
Mood | Change from Baseline Mood at 2 months
  Beck Depression Inventory: Individuals' emotional states were evaluated with the Turkish version of the Beck Depression Inventory (ref). BDI is a self-assessment scale designed to define and measure the severity of depression in healthy individuals and psychiatric patient groups. It consists of 21 items in total and each item is scored between 0-3. A total is obtained by summing the scores of all items. A high total score indicates a high severity of depression. 0-9 points = no depression, 10-16 points = mild depression, 17-29 points = moderate depression, 30 and above = severe depression
Trunk Flexibility Assesment | Change from Baseline Trunk Flexibility Assesment at 2 months
  For this test, individuals were asked to stand on a 15 cm high block, bend forward without bending their knees, and try to touch the tips of their toes. The distance between the fingertip and the block surface was measured with a tape measure and recorded in centimeters. With this test, flexibility of the lumbar region, hamstring and gastrocnemius muscles was evaluated.
Trunk Hyperextension Flexibility Assesment | Change from Baseline Trunk Hyperextension Flexibility Assesment at 2 months
  In this test, the individual stood facing the wall, keeping his pelvis and trunk in contact with the wall. For the initial value, the distance between the wall and the sternal notch was measured. After the pelvis was stabilized by the evaluator, the individual was asked to do trunk extension. The distance between the sternal notch and the wall was re-measured, subtracting the initial value from this value, and the amount of movement was recorded in centimeters.
Trunk Lateral Flexion Flexibility Assesment | Change from Baseline Trunk Lateral Flexion Flexibility Assesment at 2 months
  The test was performed standing with the arms by the body and the feet parallel to each other and the back against the wall. First, the place of the distal end of the middle finger of the right hand on the thigh was marked. Then, the subject was asked to lateral flex the trunk without taking his back away from the wall, while sliding his hand down on the thigh. At the last point reached, the place of the distal tip of the middle finger on the thigh was marked and the distance from the initial measurement point was measured. The same operations were repeated for the left side.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jago R, Jonker ML, Missaghian M, Baranowski T. Effect of 4 weeks of Pilates on the body composition of young girls. Prev Med. 2006 Mar;42(3):177-80. doi: 10.1016/j.ypmed.2005.11.010. Epub 2005 Dec 27. PMID 16376979
- [Background] Vaquero-Cristobal R, Alacid F, Esparza-Ros F, Lopez-Plaza D, Muyor JM, Lopez-Minarro PA. The effects of a reformer Pilates program on body composition and morphological characteristics in active women after a detraining period. Women Health. 2016 Oct;56(7):784-806. doi: 10.1080/03630242.2015.1118723. Epub 2015 Nov 19. PMID 26583914